CLINICAL TRIAL: NCT06009458
Title: Clinical Evaluation of Safety and Effectiveness for Acuity 200™ (Fluoroxyfocon A) Orthokeratology Contact Lens for Overnight Wear
Brief Title: Acuity 200™ (Fluoroxyfocon A) Orthokeratology Contact Lens for Overnight Wear
Acronym: Acuity200OK
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Acuity Polymers, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVDR 2022-01
Record Dates: First submitted 2023-04-06; First posted 2023-08-24 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Myopia
Keywords: orthokeratology; contact lens; Acuity; Overnight; myopia; myopic; astigmatism; astigmatic
MeSH Terms: conditions — Myopia; Astigmatism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Acuity 200™ (fluoroxyfocon A) Orthokeratology Contact Lens for Overnight Wear (Other): For the orthokeratology treatment the subjects will be instructed to wear the study lenses each night during the hours of sleep (for a minimum of 6 hours) and remove the lenses during the waking hours. The subject will be examined at 1 day, 1 week, 1 month, 3 months, 6 months, 9 months and 12 months after dispensing to evaluate the ocular physiology and the treatment effect. The target refractive error (sphere) will be plano for all subjects. All subjects enrolled at two of the investigational sites (targeted total of 40 subjects) will be evaluated for the stability of UCVA and manifest refraction throughout a single day on or following the 3 month, 6 month, or 9 month follow up visits. A post-treatment follow-up visit will be scheduled 1 month following discontinuation of the study lens. When it has been determined that no additional follow up visits are required, the subject will be discharged from the study.
  Interventions: Device: Acuity 200™ (fluoroxyfocon A) Orthokeratology Contact Lens for Overnight Wear

INTERVENTIONS:
Device: Acuity 200™ (fluoroxyfocon A) Orthokeratology Contact Lens for Overnight Wear — Acuity 200™ Orthokeratology Contact Lenses are intended to be worn overnight with removal during following day. The lenses are designed to produce a temporary reduction of myopia by reversibly altering the curvature of the cornea. The lenses are manufactured from fluoroxyfocon A, which is a gas permeable contact lens material composed of a siloxanyl fluoromethacrylate copolymer. The material name fluoroxyfocon A is registered with United States Adopted Name (USAN).The Acuity 200™ (fluoroxyfocon A) Orthokeratology Contact Lens is available in spherical, asymmetrical, aspheric, and tangential lens designs to best fit the individual cornea, using corneal topography and/or diagnostic lenses.

SUMMARY:
The objective of this clinical investigation is to collect scientifically valid safety and effectiveness data on the Acuity 200™ (fluoroxyfocon A) Orthokeratology Contact Lens for Overnight Wear. The clinical performance data reported from this study is intended to be submitted to the U.S. Food and Drug Administration Center for Devices and Radiological Health (CDRH) in support of a new Premarket Application (PMA).

DETAILED DESCRIPTION:
Orthokeratology is an alternative method to correct refractive errors using individually designed gas permeable (rigid) lenses worn overnight to temporarily modify the curvature of cornea. Modern orthokeratology technology uses highly permeable rigid lens material and dynamic reverse geometry designs to allow faster and more effective corneal reshaping. Acuity 200™ (fluoroxyfocon A) is a stable material with relatively higher oxygen permeability compared to other marketed gas permeable materials. The clinical effects of wearing contact lenses that limit oxygen supply have been extensively reported with potential complications related to hypoxia including corneal swelling, epithelial microcysts, limbal hyperemia, corneal vascularization, refractive error changes and corneal distortion. Given the significantly higher oxygen permeability characteristics of Acuity 200™ (fluoroxyfocon A) relative to currently FDA approved orthokeratology materials, the material is well-suited for overnight wear applications-such as orthokeratology, when the eye is subject to hypoxic conditions during sleep.

The objective of the clinical investigation (AVDR 2022-01) is to collect scientifically valid safety and effectiveness data on the Acuity 200™ (fluoroxyfocon A) Orthokeratology Contact Lens for Overnight Wear. The clinical performance data reported from the study is intended to be submitted to the U.S. Food and Drug Administration Center for Devices and Radiological Health (CDRH) in support of a new Premarket Application (PMA). The hypothesis is that the primary and secondary outcomes for safety and effectiveness are consistent with currently marketed devices approved by the FDA for overnight orthokeratology.

ELIGIBILITY:
Inclusion Criteria:

1. Is age 7 or older with full legal capacity to volunteer or has parental or legal guardian written approval to volunteer; and has read, understood and signed the Informed Consent Form or Assent Form (for subjects 18 years and under);
2. Is willing and able to follow participant instructions for product usage and meet the specified schedule of follow-up visits;
3. Has naturally occurring refractive myopia from -0.75 to -6.00 diopters sphere (spectacle plane), with refractive astigmatism (spectacle plane) up to 1.75 DC-as determined by adjusted manifest refraction (phoropter or trial frame) with a 12.5 mm vertex distance.
4. Has a best spectacle corrected visual acuity of 0.04 log MAR (20/20 -2) or better in each eye;
5. Is free of eye disease and binocular vision problems (e.g., strabismus, amblyopia, oculomotor nerve palsies, corneal disease, etc.) that may affect vision or contact lens wear; Has normal healthy eyes with no evidence of lid infection or structural abnormality; a conjunctiva free of infection; a cornea clear and free of edema, visually or topographically significant scars, clinically significant staining, significant vascularization, infiltrates when examined by slit-lamp biomicroscopy; and no evidence of iritis or uveitis.

Exclusion Criteria:

1. Is pregnant, breast-feeding or intends to become pregnant over the course of the study.
2. Is a potential pediatric subject that does not have the appropriate level of psychological maturity to comply with appropriate procedures needed for safe wear according to the investigator.
3. Is a potential pediatric subject that is a ward of the State or any other agency, institution, or entity.
4. Has a history of any of the following medical conditions: collagen vascular disease, autoimmune disease, immunodeficiency diseases, ocular herpes zoster or simplex, endocrine disorders (including, but not limited to active thyroid disorders and diabetes), lupus, and rheumatoid arthritis. NOTE: The presence of diabetes (either type 1 or 2), regardless of disease duration, severity or control, specifically excludes subjects from eligibility.
5. Has a history of intraocular or corneal surgery (including cataract extraction and refractive surgery-such as Lasik), active ophthalmic disease or abnormality (including, but not limited to, blepharitis, recurrent corneal erosion, dry eye syndrome, neovascularization > 1mm from limbus), clinically significant lens opacity, clinical evidence of trauma (including scarring), or with evidence of glaucoma or propensity for narrow angle glaucoma as determined by gonioscopic examination in either eye. NOTE: This includes any subject with open angle glaucoma, regardless of medication regimen or control. Additionally, any subject with an IOP greater than 21 mm Hg at baseline is specifically excluded from eligibility.
6. Has evidence of keratoconus, corneal irregularity, or abnormal video-keratography in either eye.
7. Has a pupil size greater than 6.0 mm in photopic illumination as measured with pupil detection component of computer assisted video keratography.
8. Has a corneal diameter of 10 mm or less;
9. Has flat keratometry values flatter than 38.00D (8.88 mm), or steeper than 47.00D (7.16 mm);
10. Takes medication that may cause dry eye or affect vision, corneal curvature, or healing (i.e., corticosteroids);
11. Has an allergy to any ingredient in the study lens care solutions;
12. Has significant ocular allergy, which would contraindicate solution use and/or "normal" contact lens wear;
13. Is currently using or has a history of atropine use for myopia progression control
14. Is a current wearer or previous wearer within the last 90 days of daily wear rigid gas permeable contact lenses, extended wear rigid gas permeable contact lenses, or orthokeratology contact lenses;
15. Is participating in any other type of clinical or research study.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 387 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Lines of improvement of monocular UCVA at the 12-month visit (overall and stratified by baseline sphere) | 1 year
  The number of lines of change in acuity (for an eye) is defined as the difference in the logMAR acuities, scored to the letter, multiplied by 10. Each line difference represents 0.1 logMAR acuity. The improvement in acuity is represented by a numerical reduction in the logMAR value.
  The primary effectiveness endpoints described above will also be stratified by subjects' baseline age (including 7 to 11 years (children), 12 to 21 years (adolescents), and 22 years and older (adults) .
Attempted vs. Achieved Reduction in manifest refractive error | 1 Year
  proportion of eyes with manifest sphere within ±0.50 D, ±1.00 D, and ±2.00 D of the target (plano) at the 12-month post-dispensing visit (overall and stratified by baseline sphere).
  The primary effectiveness endpoints described above will also be stratified by subjects' baseline age (including 7 to 11 years (children), 12 to 21 years (adolescents), and 22 years and older (adults) .
Proportion of eyes achieved UCVA of ≤0.30 logMAR , ≤0.20 logMAR ,≤0.10 logMAR, and ≤0.00 logMAR | 1 Year
  Proportion of eyes at the 1-month visit (and later visit intervals) that have achieved UCVA of ≤0.30 logMAR, ≤0.20 logMAR, ≤0.10 logMAR, and ≤0.00 logMAR for the whole cohort and stratified by pre-treatment refractive bin.
  The primary effectiveness endpoints described above will also be stratified by subjects' baseline age (including 7 to 11 years (children), 12 to 21 years (adolescents), and22 years and older (adults) .
Treatment stability | 1 Year
  Treatment stability as measured by the percentage of eyes that change by less than ±0.50 diopters manifest refraction spherical equivalent (MRSE) between two consecutive visits (baseline and 1-month, 1 and 3-month, 3 and 6-month, 6 and 9-month, and 9 and 12-month)
  The primary effectiveness endpoints described above will also be stratified by subjects' baseline age (including 7 to 11 years (children), 12 to 21 years (adolescents), and 22 years and older (adults) .
Number and rates (by type of event and relation to device) of serious and significant adverse events occurred at any visit | 1 Year
  Number and rates (by type of event and relation to device) of serious and significant adverse events occurred at any visit.
  The primary safety endpoints described above will also be stratified by subjects' baseline age (including 7 to 11 years (children), 12 to 21 years (adolescents), and 22 years and older (adults).
Number and rates (by type of event) of all types of adverse events that were not classified as serious or significant adverse events. | 1 Year
  Number and rates (by type of event) of all types of adverse events that were not classified as serious or significant adverse events.
  The primary safety endpoints described above will also be stratified by subjects' baseline age (including 7 to 11 years (children), 12 to 21 years (adolescents), and 22 years and older (adults).
All slit lamp results will be tabulated and findings above grade 2 will be evaluated and explained in relation to the treatment | 1 Year
  All slit lamp results will be tabulated and findings above grade 2 will be evaluated and explained in relation to the treatment.
  The primary safety endpoints described above will also be stratified by subjects' baseline age (including 7 to 11 years (children), 12 to 21 years (adolescents), and 22 years and older (adults).
Number and rate of cases of loss from baseline to any post-dispensing visit of: monocular best spectacle corrected visual acuity (BSCVA) of 2 or more lines (≥ 0.2 logMar), and 1 or more lines (≥ 0.1 logMar). | 1 Year
  Number and rate of cases of loss from baseline to any post-dispensing visit of: monocular best spectacle corrected visual acuity (BSCVA) of 2 or more lines (≥ 0.2 logMar), and 1 or more lines (≥ 0.1 logMar).
  The primary safety endpoints described above will also be stratified by subjects' baseline age (including 7 to 11 years (children), 12 to 21 years (adolescents), and 22 years and older (adults).

SECONDARY OUTCOMES:
A set of descriptive statistics of improvement of monocular UCVA at all visits (1 month or later), as well as stratified by baseline sphere and by spherical equivalent. | 1 Year
  A set of descriptive statistics of improvement of monocular UCVA at all visits (1 month or later), as well as stratified by baseline sphere and by spherical equivalent.
Change in best corrected spectacle visual acuity (BCSVA) from at all visits stratified by baseline pretreatment diopteric group. | 1 Year
  Change in best corrected spectacle visual acuity (BCSVA) from at all visits stratified by baseline pretreatment diopteric group.
Pre-treatment manifest sphere in comparison to post-treatment manifest sphere stratified by dioptric power for all completed subjects at the 1 month visit and later visit intervals (3, 6, 9, and 12 month visits) | 1 Year
  Pre-treatment manifest sphere in comparison to post-treatment manifest sphere stratified by dioptric power for all completed subjects at the 1 month visit and later visit intervals (3, 6, 9, and 12 month visits)
A level of attempted versus achieved reduction in manifest refractive error- proportion of eyes with manifest sphere within ±0.50 D, ±1.00 D, and ±2.00 D of the target (plano) at all other visits (1 month or later) | 1 Year
  A level of attempted versus achieved reduction in manifest refractive error- proportion of eyes with manifest sphere within ±0.50 D, ±1.00 D, and ±2.00 D of the target (plano) at all other visits (1 month or later) (overall and stratified by baseline sphere).
Corneal topography changes (in simulated keratometry flat and steep meridia) from baseline to 12-month post-dispensing visit (overall and stratified by baseline sphere). | 1 Year
  Corneal topography changes (in simulated keratometry flat and steep meridia) from baseline to 12-month post-dispensing visit (overall and stratified by baseline sphere).
An analysis of corneal topography for changes in eccentricity from baseline to 12-month visit | 1 Year
  An analysis of corneal topography for changes in eccentricity from baseline to 12-month visit
An analysis of change in absolute corneal astigmatism from baseline to 12-month visit | 1 Year
  An analysis of change in absolute corneal astigmatism from baseline to 12-month visit
Number of discontinued subjects and the reasons of discontinuation. | 1 Year
  Number of discontinued subjects and the reasons of discontinuation.
An analysis of the relationship between changes in simulated keratometry and corresponding reductions in manifest sphere at all scheduled visits (1 month and later). | 1 Year
  An analysis of the relationship between changes in simulated keratometry and corresponding reductions in manifest sphere at all scheduled visits (1 month and later).
Number and rates of average wear time per day at all scheduled visits (1 day and later) | 1 Year
  Number and rates of average wear time per day at all scheduled visits (1 day and later).
An analysis of the effects of wearing time on uncorrected visual acuity (UCVA) at all visits (1 month and later) | 1 Year
  An analysis of the effects of wearing time on uncorrected visual acuity (UCVA) at all visits (1 month and later).
Stability of monocular UCVA change by post-lens removal hours for the sub-group of up to 40 participants at a single day visit (at 3-month or any later visits) - stratified by baseline MRSE. | 1 Year
  Stability of monocular UCVA change by post-lens removal hours for the sub-group of up to 40 participants at a single day visit (at 3-month or any later visits) - stratified by baseline MRSE.
Stability of manifest refractive spherical equivalent (MRSE) change by post-lens removal hours for the sub-group of up to 40 participants at a single day visit (at 3-month or any later visits) - stratified by baseline MRSE. | 1 Year
  Stability of manifest refractive spherical equivalent (MRSE) change by post-lens removal hours for the sub-group of up to 40 participants at a single day visit (at 3-month or any later visits) - stratified by baseline MRSE.
Increase in corneal/refractive astigmatism of 2D or more and 1D or more post-treatment as compared to baseline | 1 Year
  Increase in corneal/refractive astigmatism of 2D or more and 1D or more post-treatment as compared to baseline.
Signs/symptoms and complications from subjective questionnaires and reported during the study | 1 Year
  Signs/symptoms and complications from subjective questionnaires and reported during the study.
Descriptive statistics of IOP (Interocular Pressure) and for percent change from baseline of IOP value will be provided at 6-month, 12-month, and post-treatment 1-month visit. | 1 Year
  Descriptive statistics of IOP (Interocular Pressure) and for percent change from baseline of IOP value will be provided at 6-month, 12-month, and post-treatment 1-month visit.
Descriptive statistics of specular microscopy measurements for percent change from baseline of specular microscopy measurements will be provided at 12-month visit | 1 Year
  Descriptive statistics of specular microscopy measurements ( Endothelial Cell Morphology Analysis (Cell density (cells/mm2), Polymegathism (CV) and Pleomorphism (percentage of hexagonal cells)) and for percent change from baseline of specular microscopy measurements will be provided at 12-month visit.
Descriptive statistics of central corneal thickness (micron) and for percent change from baseline of central corneal thickness will be provided for post-dispensing visits at 3-month, 12-month and post-treatment 1-month visits | 1 Year
  Descriptive statistics of central corneal thickness (micron) and for percent change from baseline of central corneal thickness will be provided for post-dispensing visits at 3-month, 12-month and post-treatment 1-month visits.

CONTACTS AND LOCATIONS:
Overall Officials: Mijeong Kwon Andre, MS, Study Director — Andre Vision and Device Research
Locations (13):
- United States (9):
  - Advanced Optometry of Mission Viejo, Mission Viejo, California
  - Elsa Pao, O.D. Optometrist, Oakland, California
  - Pacific Rims Optometry, San Francisco, California
  - Silicon Valley Eye Physicians, Sunnyvale, California
  - Coan Eye Care, Ocoee, Florida
  - Center for Ophthalmic and Vision Research, LLC, New York, New York
  - Reed Eye Associates, Pittsford, New York
  - Bellaire Family Eye Care, Bellaire, Texas
  - Queenston Eye Care, Houston, Texas
- Australia (3):
  - Innovative Eye Care, Adelaide
  - Custom Eyecare Newcastle, Cooks Hill
  - Eyeconic Optometry, Southport
- Rose Optometry, Hamilton, New Zealand